CLINICAL TRIAL: NCT03850496
Title: Dosing of Electrical Stimulation in Venous Insufficiency
Brief Title: DESIVI: Dosing of Electrical Stimulation in Venous Insufficiency
Acronym: DESIVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Actegy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15HH2472; 171441 (Other: IRAS Project ID); 15/LO/0620 (Other: National Research Ethics Number)
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Results first posted 2019-09-04 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Varicose Veins; Venous Stasis; Venous Insufficiency
Keywords: Venous
MeSH Terms: conditions — Varicose Veins; Varicose Ulcer; Venous Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (No Intervention): No device utilised for 6 weeks.
- Group B (Experimental): Revitive IX Neuromuscular Stimulation Device - Neuromuscular stimulation device used for 30 mins / day for 6 weeks.
  Interventions: Device: Revitive IX Neuromuscular Stimulation Device
- Group C (Experimental): Revitive IX Neuromuscular Stimulation Device - Neuromuscular stimulation device used for 60 mins / day for 6 weeks.
  Interventions: Device: Revitive IX Neuromuscular Stimulation Device

INTERVENTIONS:
Device: Revitive IX Neuromuscular Stimulation Device — Neuromuscular stimulation footplate device with a pre-programmed 30 minute varying electrical stimulation sequence.
  Arms: Group B; Group C

SUMMARY:
This study is designed to describe the difference in varicose vein outcomes found from using a neuromuscular electrical stimulation device for different amounts of time - Group A (control - no device), Group B (device for 30 mins per day) and Group C (device for 60 mins per day). The groups are assessed after 6 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients with chronic venous insufficiency who have the following are eligible for the study:

* Able to understand the study and provide meaningful written informed consent for the study.
* Willing, able, and committed to participate in the procedures for the full length of the study.
* All ethnic groups, male or female above the age of 18 years.
* Diagnosis of chronic venous insufficiency (C3-C5 CEAP Classification)
* Blood pressure currently under moderate control (< 160/100mmHg)
* No current foot ulceration

Exclusion Criteria:

Patients meeting any of the following criteria are to be excluded:

* Has an unstable condition (eg, psychiatric disorder, a recent history of substance abuse) that would affect compliance with protocol
* Pregnant
* Has a cardiac pacemaker, AICD or other implanted electrical device
* Has an Existing DVT.
* Has recent lower limb injury or lower back pain
* Has current foot ulceration or other skin ulcers
* Has any disorder that, in the opinion of the Investigator, might interfere with the conduct of the study.
* Has an ABPI < 0.8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raveena Ravikumar, MRCS, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: Yes
Available on request.
Supporting Information: Study Protocol, CSR
Time Frame: Post publication.
Access Criteria: On direct communication with researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 26 | 25 | 25
Completed | 25 | 24 | 21
Not Completed | 1 | 1 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 26 | 25 | 25 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (5) | 59 (5) | 63 (5) | 60 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 12 | 29
  Male | 18 | 16 | 13 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 26 | 25 | 25 | 76

OUTCOME MEASURES:

1. Primary Outcome: Venous Haemodynamics - Percent Change in Time Averaged Mean Velocity TAMV
Description: Assessment of change in venous flow utilising Time Averaged Mean Velocity (TAMV) (measured in cm/s), assessed as percentage change from baseline.
Time Frame: 0 and 6 weeks
Measure: Median (Inter-Quartile Range); unit: percentage change from device off
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 25 | 24 | 21
percentage change from device off
  0 weeks | 3.36 [-16.48 to 18.54] | 26.58 [6.65 to 92.32] | 39.49 [20.48 to 99.75]
  6 weeks | 0.46 [-20.81 to 12.26] | 27.83 [8.01 to 70.93] | 36.38 [6.45 to 108.80]

2. Secondary Outcome: Venous Flow Parameters - PV
Description: Assessment of change in venous flow utilising Peak Velocity (PV) (measured in cm/s), assessed as percentage change from baseline.
Time Frame: 0 and 6 weeks
Measure: Median (Inter-Quartile Range); unit: percentage change from device off
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 25 | 24 | 21
percentage change from device off
  0 Week | -4.760 [-25.84 to 12.61] | 202.7 [82.63 to 247.1] | 151.9 [111.3 to 234.7]
  6 Weeks | 3.360 [-17.91 to 15.13] | 145.8 [62.97 to 233.5] | 246.6 [84.66 to 297.5]

3. Secondary Outcome: Venous Flow Parameters - VF
Description: Assessment of change in venous flow utilising Volume Flow (VF) (measured in cc/min), assessed as percentage change from baseline.
Time Frame: 0 and 6 weeks
Measure: Median (Inter-Quartile Range); unit: percentage change from device off
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 25 | 24 | 21
percentage change from device off
  0 weeks | 5.525 [-14.76 to 22.48] | 28.81 [16.59 to 87.42] | 52.82 [16.99 to 92.54]
  6 weeks | -6.145 [-22.58 to 10.21] | 29.11 [5.768 to 84.21] | 52.82 [16.99 to 92.54]

4. Secondary Outcome: Microcirculatory Blood Flow
Description: Microcirculatory blood flow measure utilising flux arbitrary units.
Time Frame: 0 and 6 weeks.
Reporting Status: Not Posted

5. Secondary Outcome: Limb Volume
Description: Change in limb volume assessed in ml.
Time Frame: 0 and 6 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Venous Clinical Severity
Description: Clinical severity of venous disease as measured by the venous clinical severity score (VCSS). Scale measure from 0-30, with higher values indicating worse status. It is made up of 10 variables scored from 0-3
Time Frame: 0 and 6 weeks.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 25 | 24 | 21
Units on a scale
  0 weeks | 6 [4.5 to 8] | 6 [5 to 8] | 7 [4.750 to 9.250]
  6 weeks | 7 [5 to 9.5] | 5 [4 to 8] | 3 [2 to 6.5]

7. Secondary Outcome: Patient Compliance
Description: Compliance with device usage assessed with a patient completed diary.
Time Frame: 6 weeks.
Reporting Status: Not Posted

8. Secondary Outcome: Generic Quality of Life - EQ-5D-5L
Description: Quality of life as assessed by the EuroQol EQ-5D generic quality of life questionnaire. This measures from 1.00 (perfect life) to 0.00 (dead) and to negative values (worse than dead).
Time Frame: 0 and 6 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Generic Quality of Life - SF-12
Description: Quality of life as assessed by the Short Form 12 (SF-12) generic quality of life tool. Assessed at baseline and 6 weeks.
Time Frame: 0 and 6 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Generic Quality of Life - EQ-VAS
Description: Quality of life as assessed by the EuroQol Visual Analogue Scale (0-100) for generic Quality of life - EQ-VAS. Higher values better.
Time Frame: 0 and 6 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Disease Specific Quality of Life
Description: quality of life as assessed on the Aberdeen varicose vein questionnaire scale (0-100). This is a patient reported quality of life measure, which assesses symptoms of varicose veins. Higher values are worse.
Time Frame: 0 weeks and 6 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 25 | 24 | 21
units on a scale
  0 weeks | 18.62 [10.13 to 26.83] | 21.07 [16.34 to 29.47] | 21.30 [11.91 to 31.33]
  6 weeks | 19.72 [11.30 to 25.38] | 18.86 [14.99 to 28.52] | 15.01 [11.04 to 21.31]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes